CLINICAL TRIAL: NCT04349540
Title: A Prospective Non Interventional Study to Evaluate the Role of Immune and Inflammatory Response in Recipients of Allogeneic Haematopoietic Stem Cell Transplantation (SCT) Affected by Severe COVID19 Infection
Brief Title: Role of Immune and Inflammatory Response in Recipients of Allogeneic Haematopoietic Stem Cell Transplantation (SCT) Affected by Severe COVID19
Acronym: (COVID19_BMT)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20BO08
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: COVID19
Keywords: HSCT
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
COVID19 pandemic currently represents a public health emergency. Based on current data, 15% of the affected individuals will develop a severe form of the disease requiring admission to hospital and respiratory support. Data show that age and cardiovascular pre-existing comorbidities predict a poorer outcome. Some evidence suggests that a subset of patients with poorer outcome present with a cytokine mediated inflammatory response and with a secondary HLH like clinical phenotype. No data are so far available with regard to the risk of severe COVID19 disease in the post stem cell transplantation setting. Recipients of allogeneic stem cell transplantation are by definition immunologically dysregulated and could potentially present with a unique immune-inflammatory response to COVID 19 infection. Moreover, the immunosuppression used to prevent/treat GVHD may also impact clinical progression and it is possible that because of their immunological defects, SCT patients could potentially have prolonged carriage of the virus and hence act as "super spreaders".

The present study aims at documenting clinical and biological characteristics, including immunological profiling, of allogeneic stem cell transplant recipients presenting with severe COVID 19 infection and its impact on patients survival. This work may provide the scientific basis for targeted therapy with biological agents in this patient group.

DETAILED DESCRIPTION:
The transplant teams in each participating site will be identifying and approaching eligible patients. Adult and paediatric patients with a history of allogeneic stem cell transplantation who are admitted to hospital with a proven severe COVID19 infection will be eligible for the study. Within 72 hrs of admission, a 10 ml clotted blood (5 mls for pts below 15 kg weight) will be collected and serum frozen at -80 C. This sample will be sent with a 10ml blood sample (5 mls for pts below 15 kg weight) in EDTA to the Immunology Laboratories at Great Ormond Street Hospital (GOSH) in London for centralized cytokine and lymphocyte subset analysis. The sample will be divided into 2 aliquots, one being analyzed directly, the second one being frozen for further assays as developed. Other immunological and biochemical parameters will be tested locally and results with local reference ranges will be collected for the purpose of the current study.

In case the patient deteriorates further from the respiratory perspective requiring either CPAP or mechanical ventilation, a second 5 ml serum sample may be collected, frozen at -80 C and sent to GOSH for repeated cytokine analysis.

HScore will be calculated as per published data but bone marrow aspiration will be optional in calculating the scoring given the expected acute clinical situation of the patient. (Fardet et al, Arthritis Rheumatol 2014).

Transplant research team members will collect demographic and clinical characteristics at the time samples are sent to GOS. Blood results, data on clinical course, therapy (including biological agents) and outcome data will be collected with a follow up survey 30 and 100 days after start of supplemental oxygen therapy for COVID19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Adult and paediatric patents (any age) who have received allogeneic stem cell transplantation AND
2. Proven COVID19 infection as documented by PCR testing of nasal/ throat swab or NPA AND
3. Severe COVID 19 infection as defined by need for supplemental oxygen

Exclusion Criteria:

1. Patients beyond the first 72 hours of developing oxygen requirement or
2. Patients who have received cytokine targeting treatment before blood sampling or
3. Patients with a mild/moderate COVID19 infection (ie no need for supplementary oxygen)

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patinets who develop severe COVID19 infection (defined as requiring oxygen support) after having received an allogeneic stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of inflammatory/immunological biomarkers <72 hours after development of oxygen requirement | 72 hrs

SECONDARY OUTCOMES:
Overall survival at 30 and 100 days after development of oxygen requirement | day +30 and +100
Comparison of 30 and 100 day survival in SCT patients who are vs are not ongoing immunosuppression | Day +30 and +100
Proportion of patients requiring mechanical ventilation | Day +30
Incidence of secondary HLH (as defined by HS score) | Day +30

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No